CLINICAL TRIAL: NCT01084798
Title: A Retrospective Study On The Management of Multiple Sclerosis (MS) Over The Last 10 Years
Brief Title: A Retrospective Study to Understand the Clinical Management of Subjects With Multiple Sclerosis at a Site in Taiwan Over the Last 10 Years
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Yu-Li Wu, Attending Physician, Chang-Gung Memorial Hospital
Other Study IDs: EMR 200077-503
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2010-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Expanded Disability Status Scale; Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, non comparative, non-randomised, open-label, retrospective, single centre study planned to collect the data of subjects diagnosed with multiple sclerosis (MS) as per Poser or McDonald criteria between 1997 and 2007 in Taiwan. The clinical features and annual relapse rate in the first five years after the onset of disease have been compared between conventional and optico-spinal MS in the earlier studies. This study aims to understand the clinical care pathway of MS subjects and facilitate the subject's diagnosis before converting to MS.

DETAILED DESCRIPTION:
Multiple Sclerosis is a chronic, inflammatory disease of the central nervous system (CNS) and is characterised by areas of demyelination, or plaques in the CNS. The disease is twice as prevalent in women as compared to men and causes considerable disability over time and continues for the lifetime of the subject. Subjects with MS are thought to have a genetic predisposition for the disease, though environmental factors such as geographic location and possibly viral infection also play an important role in the process of development of the disease.

OBJECTIVES

Primary objective:

* To understand the clinical care pathways of MS subjects at the site over the last 10 years in order to raise the medical attention of MS diagnosis

Secondary objective:

* To review the pattern of MS treatment regimens in MS subjects at a particular site between 1997 and 2007

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with MS as per Poser or McDonald criteria between 1997 and 2007
* EDSS before treatment was available if subject has started the disease modifying drug treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with MS between 1997 and 2007 in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Distribution of locations (medical centre, regional hospital, general practitioners) where subjects were treated for the first episode of attack prior to multiple sclerosis diagnosis | Data collected for last 10 years between 1997 and 2007

SECONDARY OUTCOMES:
Duration from first attack to confirmation of MS | Data collected for last 10 years between 1997 and 2007
Distribution of MS diagnosis criteria and treatment regimens | Data collected for last 10 years between 1997 and 2007
Annual relapse rate before and after MS treatment | Data collected for last 10 years between 1997 and 2007
Changes in Expanded Disability Status Scale (EDSS) before and after treatment | Data collected for last 10 years between 1997 and 2007
Changes in VEP before and after treatment | Data collected for last 10 years between 1997 and 2007
Association between baseline demographics/disease characteristics and MS | Data collected for last 10 years between 1997 and 2007

CONTACTS AND LOCATIONS:
Locations (1):
- Chang-Gung Memorial Hospital, Taoyuan, Taiwan